CLINICAL TRIAL: NCT00450476
Title: Aspiration of Subglottic Secretions in Intubated Critically Ill Patients Using Hi-Lo Evac Endotracheal Tube: Correlation Between Tube Size and Incidence of Suction Lumen Dysfunction
Brief Title: Aspiration of Subglottic Secretions Using Hi-Lo Evac Endotracheal Tube: Tube Size and Incidence of Suction Lumen Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Alexandroupolis (Other)
Other Study IDs: 30/3/25-01-2007
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Aspiration of Subglottic Secretions
Keywords: ventilator associated pneumonia; prevention; endotracheal intubation; mechanical ventilation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hi-Lo Evac Endotracheal Tube

SUMMARY:
To evaluate the correlation between endotracheal tube size and incidence of dysfunction of suction lumen of Hi-Lo Evac endotracheal tube in critically ill patients who required mechanical ventilation for more than 48 hours.

DETAILED DESCRIPTION:
In mechanically ventilated patients, aspiration of subglottic secretions is a widely used intervention for prevention of ventilator-associated pneumonia. Using Hi-Lo® Evac endotracheal tube (Hi-Lo Evac; Mallinckrodt; Athlone, Ireland), dysfunction of suction lumen and subsequent failure to aspirate the subglottic secretions is not uncommon. The objective of this prospective observational study is to determine the causes and the incidence of suction lumen dysfunction of Evac endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with orotracheal intubation and anticipated duration of intubation more than 48 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Christos K Dragoumanis, MD, PhD, Principal Investigator — Intensive Care Unit, University Hospital of Alexandroupolis
Locations (1):
- University General Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece